CLINICAL TRIAL: NCT05198960
Title: AVAJAK: Apixaban/Rivaroxaban Versus Aspirin for Primary Prevention of Thrombo-embolic Complications in JAK2V617F-positive Myeloproliferative Neoplasms
Acronym: AVAJAK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC20.0263 (AVAJAK)
Record Dates: First submitted 2021-11-09; First posted 2022-01-20 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia; Prefibrotic/Early Primary Myelofibrosis; JAK2 V617F; High-risk Patients
Keywords: Venous ThromboEmbolism; Arterial Thrombosis; Hemorrhage
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Venous Thromboembolism; Hemorrhage | interventions — N(4)-oleylcytosine arabinoside; Aspirin

STUDY DESIGN:
Intervention Model Description: AVAJAK is an academic multicenter phase 3 prospective, randomized, and open label trial.
  > Randomization of the patients: Patients corresponding to inclusion criteria will be randomized based on a 1:1 distribution.
  * Experimental group (Patients allocated to receive low-dose DOAC, at the choice of the investigator)
    * Apixaban 2.5 mg BID or
    * Rivaroxaban 10 mg OD, at the choice of the investigator.
  * Control group (Patients allocated to receive LDA)
    - Aspirin 100 mg OD Dispensation of treatments every 6 months for 24 months
  * Stratification:
    * First stratification will be done by center
    * Second stratification will be done by pathology (PV/ET/ PreMF)
    * No stratification will be made based on DOAC drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients randomized to receive Direct Oral Anticoagulants, at the choice of the investigator Apixaban 2.5 mg both in day or Rivaroxaban 10 mg one per day, at the choice of the investigator
  Interventions: Drug: Direct Oral Anticoagulants
- Control group (Active Comparator): Patients randomized to receive Low-Dose Aspirin Aspirin 100 mg one per day
  Interventions: Drug: Low-dose aspirin

INTERVENTIONS:
Drug: Direct Oral Anticoagulants — Patients randomized to receive DOAC, at the choice of the investigator: Apixaban 2.5 mg both in day or Rivaroxaban 10 mg once daily.
  Arms: Experimental group
Drug: Low-dose aspirin — Patients allocated to receive LDA: Aspirin 100 mg OD once daily.
  Arms: Control group

SUMMARY:
Philadelphia-negative myeloproliferative neoplasms (MPN) are frequent and chronic myeloid malignancies including Polycythemia Vera (PV), essential thrombocythemia (ET), Primary Myelofibrosis (PMF) and Prefibrotic myelofibrosis (PreMF). These MPNs are caused by the acquisition of mutations affecting activation/proliferation pathways in hematopoietic stem cells. The principal mutations are JAK2V617F, calreticulin (CALR exon 9) and MPL W515. ET or MFP/PreMF patients who do not carry one of these three mutations are declared as triple-negative (3NEG) cases even if they are real MPN cases.

These diseases are at high risk of thrombo-embolic complications and with high morbidity/mortality. This risk varies from 4 to 30% depending on MPN subtype and mutational status.

In terms of therapy, all patients with MPNs should also take daily low-dose aspirin (LDA) as first antithrombotic drug, which is particularly efficient to reduce arterial but not venous events.

Despite the association of a cytoreductive drug and LDA, thromboses still occur in 5-8% patients/year.

All these situations have been explored in biological or clinical assays. All of them could increase the bleeding risk. We should look at different ways to reduce the thrombotic incidence: Direct Oral Anticoagulants (DOAC)? In the general population, in medical or surgical contexts, DOACs have demonstrated their efficiency to prevent or cure most of the venous or arterial thrombotic events.

At the present time, DOAC can be used in cancer populations according to International Society on Thrombosis and Haemostasis (ISTH) recommendations, except in patients with cancer at high bleeding risk (gastro-intestinal or genito-urinary cancers). Unfortunately, in trials evaluating DOAC in cancer patients, most patients have solid rather than hematologic cancers (generally less than 10% of the patients, mostly lymphoma or myeloma).

In cancer patients, DOAC are also highly efficient to reduce the incidence of thrombosis (-30 to 60%), but patients are exposed to a higher hemorrhagic risk, especially in digestive cancer patients.

In the cancer population, pathophysiology of both thrombotic and hemorrhagic events may be quite different between solid cancers and MPN. If MPN patients are also considered to be cancer patients in many countries, the pathophysiology of thrombosis is quite specific (hyperviscosity, platelet abnormalities, clonality, specific cytokines…) and they are exposed to a lower risk of digestive hemorrhages. It is thus difficult to extend findings from the "general cancer population" to MPN patients.

Unfortunately, only scarce, retrospective data regarding the use of DOAC in MPNs are available data.

We were the first to publish a "real-life" study about the use, the impact, and the risks in this population. In this local retrospective study, 25 patients with MPN were treated with DOAC for a median time of 2.1 years. We observed only one thrombosis (4%) and three major hemorrhages (12%, after trauma or unprepared surgery). Furthermore, we have compared the benefit/risk balance compared to patients treated with LDA without difference.

With the increasing evidences of efficacy and tolerance of DOAC in large cohorts of patients including cancer patients, with their proven efficacy on prevention of both arterial and venous thrombotic events and because of the absence of prospective trial using these drugs in MPN patients, we propose to study their potential benefit as primary thrombotic prevention in MPN.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of PV or ET or PreMF according to WHO or BSCH criteria (bone marrow biopsy not compulsory).
* Patients with JAK2V617F mutation (threshold allele burden > 1%).
* Patients considered as "high-risk" patients:

  1. based on age (> 60-year-old)
  2. based on thrombotic history (compatible with antithrombotic randomization) but aged ≥ 18-year-old.
* Length of time from MPN diagnostic to inclusion will not exceed 12 months.

Exclusion Criteria:

* Contra-indication to aspirin or DOAC due to allergic situation or recent history of major bleeding.
* Formal indication of treatment with aspirin or DOAC (thus precluding randomization).
* Inability to give informed consent.
* Patients under curatorship/guardianship
* Concomitant use of a strong inhibitor or inducer of CYP3A4 (like ruxolitinib).
* Chronic liver disease or chronic hepatitis.
* Renal insufficiency with creatinine <30 ml/mn on Cockcroft and Gault Formula
* Patient considered at high-risk of bleeding: patients with current or recent major or clinical relevant non major bleeding gastrointestinal or cerebral bleedings
* Planned pregnancy within 24 months
* No appropriate contraception (estrogen contraception or no contraception) in women of childbearing age or breastfeeding woman
* PS>2 or life expectancy <12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1308 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2027-07-13 (Estimated); Study Completion 2027-07-13 (Estimated)

PRIMARY OUTCOMES:
Time to occurrence of arterial or venous thromboembolic events. | Time to occurrence up to 24 months of patient follow-up
  Nb and type of thrombotic events during the FU

SECONDARY OUTCOMES:
Time to occurrence of major and clinically relevant non-major bleedings as defined by International Society on Thrombosis and Haemostasis | Time to occurrence up to 24 months of patient follow-up
  Nb and type of new hemorrhagic events
Time to occurrence of arterial thromboembolic events. | Time to occurrence up to 24 months of patient follow-up
  Nb and type of new arterial events
Time to occurrence of venous thromboembolic | Time to occurrence up to 24 months of patient follow-up
  Nb and type of new venous events
Time to occurrence of thromboembolic and bleeding events according to the cytoreductive associated drugs | Time to occurrence up to 24 months of patient follow-up
  Nb and type of new thromboembolic and hemorrhage events
Time to occurrence of serious adverse events others than thromboses and hemorrhages hemorrhages | Time to occurrence up to 24 months of patient follow-up
  Nb, type and grade of adverse events observed
Overall survival and event-free survival | 24 months
  Time to last news and time to first event
Therapeutic adherence | 24 months
  Therapeutic adherence by Girerd auto-questionnaire
Occurrence of atrial fibrillation episode (time to occurrence). | 24 months
  Nb and timing of atrial fibrillation event
Evaluation of Quality of life under antithrombotic drugs | 24 months
  Evaluation of QoL by the use of MPN-SAF Quality of life
Evaluation of costs and incremental cost utility ratio of low-dose DOAC compared to low-dose aspirin | 24 months
  Evaluation of benefits/costs under antithrombotic drugs
Evaluation of Quality of life under antithrombotic drugs | 24 months
  Evaluation of QoL by the use of EQ-5D-5L Quality of life

CONTACTS AND LOCATIONS:
Locations (42):
- France (42):
  - CHU d'Angers, Angers
  - CH d'Annecy, Annecy
  - CH d'Argenteuil, Argenteuil
  - CH d'Avignon, Avignon
  - CH de la Côte Basque Bayonne, Bayonne
  - CH de Béziers, Béziers
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - Hôpital privé Cesson-Sévigné, Cesson-Sévigné
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor (APHP), Créteil
  - CHU Grenoble Alpes, Grenoble
  - CHD Vendée La Roche Sur Yon, La Roche-sur-Yon
  - CHU Le Havre, Le Havre
  - CH Le Mans, Le Mans
  - CH Libourne, Libourne
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Léon Bérard Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - CH de Morlaix, Morlaix
  - CHU de Nancy, Nancy
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - Hôpital Privé du Confluent Nantes, Nantes
  - CHR d'Orléans, Orléans
  - Hôpital St-Louis (APHP), Paris
  - Hôpital Cochin (APHP), Paris
  - CH de Perpignan, Perpignan
  - CH de Périgueux, Périgueux
  - CHIC de Quimper, Quimper
  - CHU de Rennes, Rennes
  - CH de Rochefort, Rochefort
  - CH de Roubaix, Roubaix
  - Centre Henri Becquerel de Rouen, Rouen
  - CHU La Réunion - Site Nord Félix GUYON, Saint-Denis
  - CHU La Réunion - Site Sud, Saint-Pierre
  - Institut de Cancérologie Lucien Neuwirth St-Priest-en-Jarez, Saint-Priest-en-Jarez
  - Clinique Sainte Anne Strasbourg, Strasbourg
  - CHU de Tours, Tours
  - CH Bretagne Atlantique Vannes, Vannes
  - CH de Versailles, Versailles
  - CH Paul-Brousse (APHP), Villejuif
  - Médipôle Hôpital Mutualiste Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.